CLINICAL TRIAL: NCT06223126
Title: Effects of Oral Contraceptive on Stress Reactivity and Mood Homeostasis
Brief Title: Stress Reactivity and Hormonal Contraception
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Uppsala University (Other); German Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: TUE011_IRTG_P03
Record Dates: First submitted 2024-01-15; First posted 2024-01-25 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-08

CONDITIONS: Hormonal Contraception
Keywords: Stress reactivity; Mood homeostasis; fMRI; Oral Contraceptive; Sex hormones; Cortisol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Oral Contraception-Starter: Women who start taking oral contraception
  Interventions: Other: Combined oral contraception
- Oral Contraception-Stopper: Women who stop taking oral contraception
  Interventions: Other: Discontinuation of a combined oral contraception
- Oral Contraception-Long-Term User: Women who use oral contraception continuously

INTERVENTIONS:
Other: Combined oral contraception — Women, who want to start taking birth control pills will get a prescription for oral contraception at the discretion of their own attending physician
  Groups: Oral Contraception-Starter
Other: Discontinuation of a combined oral contraception — Cessation of the use of combined oral contraceptives
  Groups: Oral Contraception-Stopper

SUMMARY:
For almost 60 years, millions of women globally have relied on oral contraceptive (OC) pills for pregnancy prevention and addressing menstrual irregularities. However, 4-10% of users experience mood-related side effects such as depression and anxiety, often leading to discontinuation of OC use. Previous studies also indicate that OC usage may lead to chronic alterations in brain structure and the regulation of the hypothalamic-pituitary-adrenal axis, a system involved in regulating stress responses. In the proposed study the investigators aim to investigate in more detail how women who start taking oral contraception (OC) and women who stop taking OC differ in their stress reactivity and their mood from long-term OC users. Furthermore, assessing hormones will help to shed light on the connection between OC, stress reaction, sex hormones and the brain. To achieve this, individual biomarkers will be evaluated, including changes in brain anatomy, functional responses and connectivity during acute psychosocial stress and early changes in mood and well-being through ambulatory assessment.

DETAILED DESCRIPTION:
The study will use a longitudinal design with two time points to compare three groups, the women who want to start taking the pill, the women who want to stop taking it, and those who are long-term users of the pill. They will be exposed to a psychosocial stress induction task (Montreal Imaging Stress Task; MIST) in functional magnetic resonance imaging (fMRI) to get mechanistic insights. Measurements will be done before and during OC use (group 1; OC-Starters) and during and after the termination of OC use (group 2; OC-Stoppers). Therefore, at the first time point (T1) of the measurements, the OC-Starter will be in their early follicular phase while the OC-Stopper will be in their active pill intake weeks. At the second time point (T2), the OC-Starter will be in the active pill intake weeks and the OC-Stopper in their early follicular phase. The OC-Long-Term users (group 3) will be in their active pill intake weeks at both measurement time points (T1 and T2). Along with measuring heart rate, skin conductance and pulse oximetry as indicators of stress, saliva samples will be collected during the assessment in the fMRI to determine cortisol levels. Hormones (e.g., estradiol, ethinylestradiol, testosterone, and their precursor steroids and metabolites) will be assessed from blood samples at both time points (T1 and T2). Hair samples are collected at both measurement time points (T1 and T2) from the study participant to record the cumulative cortisol secretion of the past 3 months (= 3cm of hair) as a marker for chronic stress. For this purpose, a small strand of hair on the back of the head of the participant will be cut as close to the scalp as possible. These measures will be analyzed alongside individual markers of stress responsivity derived from brain imaging and questionnaires on stress and emotion regulation. These trait-like measures will be assessed at baseline (T1) and three months after the start/end of OC use (T2) to evaluate long-term changes. Additionally, at T1 and T2, medically trained personnel will conduct transvaginal ultrasound examinations to visualize the female reproductive organs and assess any organic changes resulting from OC usage. After the first time point T1, ambulatory assessments will be utilized over three months in all groups to assess daily fluctuations in stress and mood over the transition period starting or stopping OC and to ensure ecological validity of mood and stress reactivity. For this purpose, changes in average mood and mood variations will be quantified by collecting self-reports of daily hassles. A voluntary follow-up questionnaire is then used after six months (T3) to assess long-term changes in mood and stress reactivity.

ELIGIBILITY:
Inclusion Criteria:

* Women, who want to start using oral contraception (no hormonal contraception use for at least 4 months; regular menstrual cycle (between 25 and 35 days) prior to participation)
* Women, who want to stop using oral contraception (OC pill use for at least 6 months; regular intake of OC pill)
* Long-term oral contraception user (OC pill use for at least 6 months; regular intake of OC pill)
* German language fluency
* Normal or corrected vision
* Body-mass index (BMI): 18-35 kg/m2

Exclusion Criteria:

* Neurological or psychiatric disease
* Medical problems such as hormonal, metabolic, or chronic diseases (e.g., severe hypertension, diabetes, or congestive heart failure)
* Pregnancy, delivery, and lactation (current and within the last year)
* Any kind of steroid hormonal, pharmacological treatment, or psychotropic treatment in the last three months
* Shift work
* Participants engaging in competitive sports
* contraindication for MRI
* People with non-removable metal objects on or in the body
* Tattoos (if not MRI-incompatible according to expert guidelines)
* Pathological hearing or increased sensitivity to loud noises
* Claustrophobia
* Surgery less than three months ago
* Neurological disease or injury
* Moderate or severe head injury
* Intake of antidepressants or neuroleptics

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Stress-induced changes in mood | Pre medication vs. 3 months after medication
  Change in mood after stress inductions measured by ratings of positive and negative affect before and after the stress task will be measured with the PANAS questionnaire (scale 1-5).
  It will be measured twice three months apart; each time: 60min before stress onset, just before stress onset, immediately after stress, 40min after stress onset, 60min after stress onset, 90min after stress onset.
Stress-induced changes in the subjective experience of stress | Pre medication vs. 3 months after medication
  Change in subjective stress experience after stress inductions measured by stress items before and after the stress task will be measured with a visual analog scale (1-10).
  It will be measured twice three months apart; each time: 60min before stress onset, just before stress onset, immediately after stress, 40min after stress onset, 60min after stress onset, 90min after stress onset.
Stress-induced changes in brain response | Pre medication vs. 3 months after medication
  BOLD response to stress (changes in amplitude) within regions associated with stress reactivity and regulation (amygdala, hippocampus, prefrontal cortex, anterior cingulate cortex (ACC), middle frontal gyrus (MFG), right superior temporal gyrus (STG), insula, striatum, and praecuneus) will be quantified using fMRI to assess differences between stress vs. control conditions during the stress task.
Stress-induced changes in functional connectivity | Pre medication vs. 3 months after medication
  Functional connectivity will be assessed within regions associated with emotional processing (amygdala, hippocampus, prefrontal cortex, hypothalamus, striatum, insula) using fMRI to assess differences between stress vs. control conditions during the stress task.
Stress-induced changes in skin conductance | Pre medication vs. 3 months after medication
  Skin conductance [μS] during stress condition vs. no stress condition as indicators of stress during fMRI
Stress-induced changes in pulse | Pre medication vs. 3 months after medication
  Pulse oximetry during stress condition vs. no stress condition as indicators of stress during fMRI
Stress-induced changes in cortisol | Pre medication vs. 3 months after medication
  Salivary cortisol levels to determine cortisol levels [μg/dL or nmol/L] during stress condition vs. no stress condition and baseline as indicators of stress/Hypothalamic-Pituitary-Adrenal-axis activation.
  It will be measured twice three months apart; each time: 60min before stress onset, just before stress onset, immediately after stress, 40min after stress onset, 60min after stress onset, 90min after stress onset.
Oral Contraceptive induced changes in average mood during transition phase | Over the course of three months regularly (30 times in total), about 5 minutes per day
  Changes in positive and negative mood ratings (5 mood and 5 stress items, scale 1-10), measured with ecological momentary assessment after starting vs. stopping oral contraceptive intake.

SECONDARY OUTCOMES:
Oral Contraceptive induced changes in hormone levels | Pre medication vs. 3 months after medication
  Changes in endogenous and synthetic hormone levels will be assessed from blood samples before and after starting vs. stopping oral contraceptive use.
Oral Contraceptive induced changes in brain volume (structure) | Pre medication vs. 3 months after medication
  Changes operationalized with a structural T1 scan of the whole brain before and after starting vs. stopping oral contraceptive use.
Oral Contraceptive induced changes in chronic stress | Pre medication vs. 3 months after medication
  Associations of chronic stress, assessed via hair cortisol measures and chronic stress questionnaire (Trier Inventar of Chronic Stress - TICS; value range = [0 228]; higher outcome relates to a higher chronic stress rating) with oral contraception and stress reactivity. To record the cumulative cortisol secretion of the past 3 months (= 3cm of hair) as a marker for chronic stress, a small strand of hair on the back of the head of the participant will be cut as close to the scalp as possible.
Oral Contraceptive induced organic changes in reproductive organs | Pre medication vs. 3 months after medication
  Changes operationalized with a transvaginal ultrasound to examine the female reproductive organs (uterus, fallopian tubes and ovaries) before and after starting vs. stopping oral contraceptive use.
Oral Contraceptive induced long-term changes in mood | Six months after medication change
  Changes in positive and negative mood ratings measured with the PANAS questionnaire (scale 1-5)

CONTACTS AND LOCATIONS:
Overall Officials: Nils B. Kroemer, Professor, Principal Investigator — Department of Psychiatry & Psychotherapy, University of Tübingen
Locations (1):
- Department of Psychiatry & Psychotherapy, University of Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
After the publication of the key results of the study, all anonymized research data, including imaging data, will be made publicly available (e.g., at openfmri.org).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available after an embargo period of 12 months after completion of the study
Access Criteria: Until the data is publicly available, researchers may contact the lead PI to gain access
URL: http://neuromadlab.com